CLINICAL TRIAL: NCT03325907
Title: Transthoracic Needle Biopsy for the Diagnosis of Pulmonary Nodule Using Three-dimensional Printed Navigational Template: A Phase I Feasibility Trial
Brief Title: Transthoracic Needle Biopsy Using 3D Printed Navigational Template: A Phase I Feasibility Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Chang Chen, Prof. Dr., Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: K17-155
Record Dates: First submitted 2017-10-26; First posted 2017-10-30 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Lung Neoplasms
Keywords: Biopsy, Needle; Printing, Three-Dimensional; Image-Guided Biopsy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: single-armed feasibility trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- template-guided biopsy (Experimental): Participants receive transthoracic lung biopsy guided by navigational template.
  Interventions: Device: navigational template

INTERVENTIONS:
Device: navigational template — The navigational template was created based on computed tomography data using three-dimensional technology.

SUMMARY:
This study evaluates the feasibility of three-dimensional printed template in transthoracic pulmonary nodule biospy. Investigator planned to include 20 patients with lung nodule biopsy schedule to receive template-guided transthoracic needle aspiration.

DETAILED DESCRIPTION:
In previous study,a navigational template has been created to simplify the procedure of preoperative lung nodule localization. It was reported that localizer deviation was 10(0-20)mm.In this trial,Investigator explores the utility of this navigational template in transthoracic lung nodule biopsy.

ELIGIBILITY:
Inclusion Criteria:

CT confirmed peripheral lung nodule; Nodule size larger than or equal to 3 cm; ECOG Performance Status 0-2 ; Informed consent.

Exclusion Criteria:

Nodule located in the scapula region wherein biopsy needle is impeded; Nodule within 3 cm above diaphragmatic dome.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-08-03 (Actual); Study Completion 2020-09-03 (Actual)

PRIMARY OUTCOMES:
Success rate of needle insertion | 15 minutes
  Clinician evaluate the relative position between biopsy needle and the target lesion on CT images after needle insertion.

SECONDARY OUTCOMES:
procedural length | 1 hour
  The length of procedural time is measured from the time a patient is lying on the examining bed of the CT scanner to the time he/she complete the biopsy procedure and step off the CT table.
radiation dosage | 1 hour
  How much radiation exposure patients would receive in the whole process of transthoracic needle biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Chang Chen, MD,Ph.D, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhang L, Li M, Li Z, Kedeer X, Wang L, Fan Z, Chen C. Three-dimensional printing of navigational template in localization of pulmonary nodule: A pilot study. J Thorac Cardiovasc Surg. 2017 Dec;154(6):2113-2119.e7. doi: 10.1016/j.jtcvs.2017.08.065. Epub 2017 Sep 1. PMID 29017792
- [Derived] E H, Chen J, Sun W, Zhang Y, Ren S, Shi J, Wen Y, Su C, Ni J, Zhang L, He Y, Chen B, Casal RF, Kheir F, Ishiwata T, Zhang J, Zhao D, Chen C. Three-dimensionally printed navigational template: a promising guiding approach for lung biopsy. Transl Lung Cancer Res. 2022 Mar;11(3):393-403. doi: 10.21037/tlcr-22-172. PMID 35399565